CLINICAL TRIAL: NCT03731780
Title: Personalized Caries Management Versus Standard of Care for Preventing Incidence of Caries in Young Egyptian Adults: A Randomized Controlled Trial
Brief Title: Personalized Caries Management Versus Standard of Care for Preventing Incidence of Caries in Young Egyptian Adults
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Sherif Khadr, Doctoral Candidate, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2018cons1
Record Dates: First submitted 2018-10-31; First posted 2018-11-06 (Actual); Last update posted 2018-11-07 (Actual); Status verified 2018-11

CONDITIONS: Dental Caries
Keywords: caries, prevention, personalized medicine
MeSH Terms: conditions — Dental Caries | interventions — Chlorhexidine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: The recruiter will be blinded. The operator cannot be blinded because of the different in the procedures of caries prevention applied in each group. However, the assessors will be kept unaware of the treatment assigned to the patient.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Personalized Treatment (Experimental): Intervention by (standard preventive measures + targeting individual caries risk factors)
  Interventions: Other: Personalized Treatment
- Chlorhexidine and Rremineralization (Experimental): Intervention is (chlorhexidine + Remineralizing agent + standard preventive measures)
  Interventions: Other: Chlorhexidine and Remineralization
- Control (Active Comparator): standard preventative measures (tooth brushing, fluoride tooth paste, interdental cleaning)
  Interventions: Other: Control

INTERVENTIONS:
Other: Personalized Treatment — Targeting individual caries risk factors
  Arms: Personalized Treatment
Other: Chlorhexidine and Remineralization — chlorhexidine mouth wash and remineralizing agent
  Arms: Chlorhexidine and Rremineralization
Other: Control — Control is standard preventive measures (tooth brushing, fluoride tooth paste, interdental cleaning)
  Arms: Control

SUMMARY:
Basic standard of care emphasis only tooth brushing and flossing without addressing individual pathological factors. For this reason, randomized controlled clinical trials on personalized caries management are needed to be able to compare the effectiveness of personalized caries management to basic standard of care. This is especially true in high caries risk populations and more so for young adults who stand to benefit the most from working towards a caries free adulthood.

DETAILED DESCRIPTION:
Aim of the study: is to conduct an RCT to compare the effectiveness of a new personalized caries-control treatment protocol with standard caries treatment protocol for reducing caries incidence in high caries risk patients

Hypothesis: This project will be designed to test the null hypothesis that there is no significant difference between the new personalized caries-control treatment protocol and existing standard caries treatment protocol, and to test the alternative hypothesis that the new personalized treatment protocol will be superior to the standard preventive measures

Primary objective: is to measure the incidence of new caries lesions

ELIGIBILITY:
Inclusion Criteria:

1. High caries risk patients
2. 18-25 years
3. Males or Females
4. Patients approving to participate in the study -

Exclusion Criteria:

* Patients with systemic conditions
* Current periodontitis (sites of probing pocket depth ≥ 5 mm)
* Allergy to any of the ingredients of the study products
* Evidence of parafunctional habits
* Dysfunction of temporomandibular joint
* Use of antibiotics in the previous 30 days
* Patients with developmental dental anomalies
* Patients with removable prosthesis
* Patients with Orthodontic appliance
* Periapical Abscess or Fistula and exposed pulps.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 81 (Estimated)
Dates: Start 2018-12 (Estimated); Primary Completion 2020-03 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
incidence of new caries lesions | 12 month
  incidence of new caries lesions

CONTACTS AND LOCATIONS:
Overall Officials: Fawzi, PhD, Study Chair — Cairo University
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Data will be made available after publication upon request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 12 month after publication , data will be available upon request
Access Criteria: principal investigator to be contacted by email for data access